CLINICAL TRIAL: NCT02045056
Title: Modulation of Micro-RNA Pathways by Gemfibrozil in Predementia Alzheimer Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Gregory Jicha, 323-5550 (Other)
Responsible Party: Sponsor-Investigator, Gregory Jicha, 323-5550, Sponsor/PI, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R01AG042419 (NIH)
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Preclinical Alzheimer's Disease
Keywords: Alzheimer disease; mild cognitive impairment; normal cognition
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Gemfibrozil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemfibrozil (Experimental): Gemfibrozil 600 mg by mouth twice daily for 48 weeks
  Interventions: Drug: Gemfibrozil
- Sugar pill (Placebo Comparator): Matching placebo capsule by mouth twice daily for 48 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gemfibrozil
  Arms: Gemfibrozil
Drug: Placebo
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to assess the safety and efficacy of gemfibrozil in modulating microRNA-107 levels for the prevention of Alzheimer's disease in subjects with intact cognition and mild cognitive impairment

DETAILED DESCRIPTION:
Double-blind, placebo controlled, parallel-design. 48 cognitively-intact subjects, and 24 subjects with early cognitive decline (CDR 0.5) will be randomly assigned to treatment with gemfibrozil (600 mg orally twice a day) or placebo for 52 weeks. Safety assessments will include routine assessment of adverse events, safety labs, and brain magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following inclusion criteria in order to participate in the study:

1. Men or women aged 65-90, inclusive.
2. Stable medical condition for three months prior to screening visit, with no clinically significant abnormalities of hepatic, renal, and hematologic function defined as follows: Platelets > 100,000, Serum creatinine ≤ 1.6 mg/dL, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 1.5 upper limit of normal, No clinically significant abnormalities of other laboratory studies (CBC, chemistry panel)
3. Non-diabetic or well controlled diabetes confirmed by fasting serum glucose <126 mg/dL.
4. Stable medications for 4 weeks prior to screening visit.
5. Physically acceptable for this study as confirmed by medical history, physical exam, neurological exam and clinical tests.

   * Exceptions to these criteria may be considered on a case-by-case basis, at the discretion of the Project Director.

Exclusion Criteria:

1. Female participants that are pregnant or of childbearing potential.
2. Unstable medical conditions for three months prior to screening visit such as poorly controlled blood pressure, diabetes, or breathing problems…etc.
3. Clinically significant abnormalities on liver, kidney or other blood tests
4. Significant neurologic disease such as Alzheimer's disease, Parkinson's disease, stroke, brain tumor, multiple sclerosis or seizure disorder.
5. Major depression in past 12 months (DSM-IV criteria), major mental illness such as schizophrenia, or recent (in past 12 months) alcohol or substance abuse.
6. History of invasive cancer within the past two years.
7. Contra-indications to lumbar puncture (bleeding disorder, platelet count < 100,000, anticoagulant treatment, major structural abnormality or sepsis in the area of the lumbosacral spine that would make a lumbar puncture technically difficult).
8. Use of any investigational agents within 30 days prior to screening.
9. Contra-indications to MRI (metallic implants, pacemaker, shrapnel, ect…)
10. Sensitivity, intolerance, or allergies to gemfibrozil or any previous reaction to any cholesterol lowering medicine.
11. Major surgery within eight weeks prior to the Baseline Visit.
12. Blindness, deafness, language difficulties or any other disability which may prevent the potential participant from participating or cooperating in the protocol.
13. Physically unacceptable for this study as confirmed by medical history, physical exam, neurological exam and clinical tests.

    * Exceptions to these criteria may be considered on a case-by-case basis, at the discretion of the examining study physician.

Excluded Medications:

1. Experimental drugs
2. Repaglinide
3. "Statins" including but not limited to atorvastatin (Lipitor), fluvastatin (Lescol), lovastatin (Mevacor), pravastatin (Pravachol), rosuvastatin (Crestor), simvastatin (Zocor), or any combination medicines containing these drugs.
4. Coumadin, warfarin, heparin, lovenox, Xarelto, apixaban or other anticoagulants. (Antiplatelet therapy is acceptable).

NOTE: If these drugs are discontinued 4 weeks or more before screening, then the participant can be eligible for the study.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Safety | 52 weeks
  Adverse events reported during the course of the trial
microRNA-107 levels | 48 weeks
  MicroRNA-107 levels will be measured in serum and cerebrospinal fluid
beta-amyloid levels | 48 weeks
  Beta-amyloid 1-40 and 1-42 levels will be measured in cerebrospinal fluid at baseline and at 48 weeks

SECONDARY OUTCOMES:
Free and cued selective reminding test (FCSRT) | 48 weeks
  The FCSRT is a sensitive measure of memory performance that will be measured at baseline and after 48 weeks of gemfibrozil treatment
Paired associates learning (PAL) | 48 weeks
  The PAL is a sensitive, computerized measure of memory performance that will be measured at baseline and after 48 weeks of gemfibrozil treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Jicha, MD, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No